CLINICAL TRIAL: NCT06864104
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Monthly Subcutaneous Administration of Tonlamarsen in Participants With Uncontrolled Hypertension (KARDINAL)
Brief Title: A Study to Investigate Tonlamarsen for the Treatment of Adults With Uncontrolled Hypertension (KARDINAL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kardigan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLA-201
Record Dates: First submitted 2025-02-12; First posted 2025-03-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Once eligibility is confirmed during screening, there will be two run-in periods (Part A and Part B). Eligible participants will then be randomized to tonlamarsen or placebo (Part C).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tonlamarsen (Experimental): 1 dose of placebo and 5 doses of active drug will be administered by subcutaneous (SC) injection
  Interventions: Drug: Tonlamarsen
- Placebo (Placebo Comparator): 5 doses of placebo and 1 dose of active drug will be administered by subcutaneous (SC) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonlamarsen — Tonlamarsen will be administered subcutaneously (SC) every 4 weeks during the randomized part of the study
  Arms: Tonlamarsen
Drug: Placebo — Placebo will be administered subcutaneously (SC) every 4 weeks during the randomized part of the study
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the blood pressure (BP)-lowering efficacy of tonlamarsen in adult participants who, despite taking 2 or more antihypertensive medications, have not achieved their target blood pressure (BP).

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 to 80, body weight ≥ 50 kg
* Has uncontrolled hypertension while receiving between 2 and 5 antihypertensive medications prescribed for hypertension
* Has mean office seated systolic blood pressure > 135 to ≤ 170 mmHg

Key Exclusion Criteria:

* Has known history of secondary hypertension
* Has documented history of poor adherence to antihypertensive medication
* Has unstable/underlying known cardiovascular disease
* Has abnormal thyroid function with clinical significance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of tonlamarsen on plasma angiotensinogen (AGT) levels | Week 20
  Percent Change from baseline (Week 0) in plasma angiotensinogen (AGT) levels to Week 20
To assess the systolic blood pressure-lowering efficacy of tonlamarsen | Week 20
  Change from baseline (Week 0) in mean office seated systolic blood pressure to Week 20

SECONDARY OUTCOMES:
To assess the safety and tolerability of tonlamarsen | Week 28
  Incidence and severity of treatment emergent adverse events (TEAEs). Incidence of clinically significant abnormalities in laboratory assessments, ECGs and vital signs. Incidence of: (1) Hyperkalemia, defined as serum potassium >5.5 mmol/L. (2) Hypotension, defined as systolic blood pressure <90 mmHg, or systolic blood pressure <100 mmHg and symptomatic and/or requiring clinical intervention. (3) Renal dysfunction, defined as a decrease of eGFR >30% from baseline value. (4) Increased proteinuria, defined as UPCR >0.5 mg/mg from baseline value.
To assess the efficacy of tonlamarsen in achieving office seated systolic blood pressure <130 mmHg | Week 20
  Proportion of participants with mean office seated systolic blood pressure <130 mmHg at Week 20
To assess the systolic blood pressure-lowering efficacy of tonlamarsen | Week 20
  Change from baseline (Week 0) in mean self-assessed home systolic blood pressure through Week 20
To assess the effect of tonlamarsen on severe systolic blood pressure elevations | Week 20
  Proportion of participants with any daily average home systolic blood pressure ≥150 mmHg at Week 20
To assess the diastolic blood pressure-lowering efficacy of tonlamarsen | Week 20
  Change from baseline (Week 0) in mean office seated diastolic blood pressure to Week 20

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Pinnacle Research Group, Anniston, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - North Coast Cardiology, Encinitas, California
  - Orange County Research Center, Lake Forest, California
  - Clinical Trials Research, Lincoln, California
  - American Institute of Research, Los Angeles, California
  - Homestead Associates in Research, Inc., Homestead, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Velocity Clinical Reseach, Savannah, Georgia
  - Eagle Clinical Research, Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Koch Family Medicine Clinical Research, Morton, Illinois
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - IMA Clinical Research, Monroe, Louisiana
  - DelRicht Clinical Research - New Orleans, New Orleans, Louisiana
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Oakland Medical Research Center, Troy, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Richmond University Medical Center, Staten Island, New York
  - CHEAR Center LLC, The Bronx, New York
  - IMA Clinical Research, Lenoir, North Carolina
  - Clinical Trials of South Carolina, Moncks Corner, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Holston Medical Group, Kingsport, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Advanced Medical Trials, LLC, Georgetown, Texas
  - Juno Research, LLC, Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - Synergy Groups Medical, LLC, Missouri City, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - Sun Research Institute, San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No